CLINICAL TRIAL: NCT04458506
Title: Treatment of Unilateral Posterior Cross Bite in the Mixed Dentition; a Randomized Controlled Trial
Brief Title: Treatment of Unilateral Posterior Cross Bite in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Region Jönköping County (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260581
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-04

CONDITIONS: Malocclusion; Maxillary Expansion; Pain Children
MeSH Terms: conditions — Malocclusion | interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Maxillary Expander (RME) (Experimental): 36 patients will be treated with RME in order to correct their unilateral posterior cross bite
  Interventions: Procedure: Maxillary expansion
- Quad Helix (QH) (Active Comparator): 36 patients will be treated with QH in order to correct their unilateral posterior cross bite
  Interventions: Procedure: Maxillary expansion

INTERVENTIONS:
Procedure: Maxillary expansion — Correction of the unilateral posterior cross bite in children

SUMMARY:
Rapid maxillary expansion and quad-helix are two well established appliances in dentistry used for posterior cross bite treatment. This study aims to compare this two different appliances in patients in their early mixed dentition, regarding treatment effects of the extra oral soft tissue but also dental and skeletal effects, if the children experience any pain and discomfort during treatment and the study also aims to make a cost minimization analysis. Comparison of these different treatments are barely made and no randomized controlled trial is yet published. No study has evaluated the difference of subjective experience during these two treatments. After this study we will know which one of these two appliances are the most effective, regarding cost minimization and treatment result but we are also able to put it in relation to the patients subjective experience

ELIGIBILITY:
Inclusion Criteria:

* Children in the early mixed dentition
* Unilateral posterior cross bite including the first permanent molar

Exclusion Criteria:

* No ongoing sucking habits
* Craniofacial syndroms
* Earlier Orthodontic treatments
* Not able to independently understand and answer the questionnaires

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Skeletal expansion at the level of the palatal median suture - the change fram Baseline | At baseline, directly after expansion and one year after expansion
  Skeletal expansion evaluated by computed tomography at three time points in both arms. The change in width of the palatal median suture is going to be evaluated and compared to the Baseline values, in both arms.
The change of inclination of teeth and alveolar bone and side effects between the time points | At baseline, directly after expansion and one year after expansion
  Dental effects and side effects evaluated by computed tomography at three time points in both arms.The change in degree of angulation and inclination of the dental structures (e.g. tooth inclinations) is going to be evaluated and compared to the Baseline values, in both arms.

SECONDARY OUTCOMES:
Assessment of the soft tissue changes | At baseline, directly after expansion, six months and one year after expansion
  3D assessment of the soft tissue changes during and after treatment by 3D -photography
Evaluation of pain and discomfort | Three times during the first week after inserting the appliances
  Questionnaire The Questionnaire has some questions with Visual Analogue Scale. With the minimum value of "0" and maximum value of "10". Higher values mean worse outcome.
  Other questions in the questionnaire have a "yes" and "No" nature.
Evaluation of Temporomandibular Disorder (TMD) | Baseline and one year after expansion
  Questionnaire The questionnaire has no scale and the questions have a "Yes" och "No" nature.
Cost-effectiveness of two treatment modalities in treatment of posterior cross bite | Through study completion, an average of 18 months
  Evaluation of both the direct and indirect costs of the treatment, number of emergency visits, treatment duration (in total) etc are going to be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Farhan Bazargani, DDS, PhD, Study Director — Örebro University, Sweden
Locations (1):
- Postgraduate Dental Education Center, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petren S, Bondemark L, Soderfeldt B. A systematic review concerning early orthodontic treatment of unilateral posterior crossbite. Angle Orthod. 2003 Oct;73(5):588-96. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 14580028
- [Derived] Hansson S, Lindsten R, Josefsson E, Birk L, Ovsenik M, Petren S, Magnuson A, Bazargani F. Three-dimensional evaluation of palatal vault changes after unilateral posterior crossbite correction with quad helix or rapid maxillary expansion: A randomized controlled trial with 1-year follow-up. Int Orthod. 2026 Jan 12;24(2S):101136. doi: 10.1016/j.ortho.2025.101136. Online ahead of print. PMID 41529457
- [Derived] Hansson S, Josefsson E, Lindsten R, Magnuson A, Bazargani F. Pain and discomfort during the first week of maxillary expansion using two different expanders: patient-reported outcomes in a randomized controlled trial. Eur J Orthod. 2023 May 31;45(3):271-280. doi: 10.1093/ejo/cjac067. PMID 36331513